CLINICAL TRIAL: NCT00410995
Title: Effects of Naproxen on Physical Performance
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never initiated.
Sponsor: University of Oklahoma (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11186
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2007-10-11 (Estimated); Status verified 2007-10

CONDITIONS: Healthy
Keywords: Physically fit volunteers
MeSH Terms: interventions — Naproxen

INTERVENTIONS:
Drug: Naproxen

SUMMARY:
The purpose of this study is to determine the effect of daily use of Naproxen (a commonly used over-the-counter NSAID) on the physical performance of athletes, as measured by maximum oxygen consumption.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or greater than18 years of age
2. No history of allergy or adverse reaction to any NSAID
3. No use of any NSAID in past 2 weeks
4. No history of peptic ulcer disease (PUD), gastroesophageal disease (GERD), or gastritis
5. No major medical history including but not limited to diabetes, hypertension, asthma, kidney disease and coronary artery disease
6. Currently not taking any medication including oral contraceptives

Exclusion Criteria:

1. Age < 18 years of age
2. History of allergy or adverse reaction to any NSAID
3. Use of any NSAID in past 2 weeks
4. History of a bleeding disorder
5. History of PUD, GERD, or gastritis
6. Pregnant
7. A medical history of diabetes, hypertension, asthma, kidney disease or coronary artery disease
8. Taking any medication including oral contraceptives

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2004-05; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Effects on physical performance in terms of maximum oxygen consumption

CONTACTS AND LOCATIONS:
Overall Officials: LaMont Cavanagh, MD, Principal Investigator — University of Oklahoma-Tulsa
Locations (1):
- Family Practice - CMT, Tulsa, Oklahoma, United States